CLINICAL TRIAL: NCT06513793
Title: The Effect of a Nature-based, Self-help Intervention on Mental Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5412277
Record Dates: First submitted 2024-07-11; First posted 2024-07-22 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Low Mental Wellbeing
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: This is a pilot randomised controlled trial with two arms; psychological intervention versus waiting list control. The control arm participants will be offered the intervention following the end of the waiting list period.
Who Masked: Outcomes Assessor
Masking Description: Outcomes are recorded remotely by the participant, online using the Qualtrics platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Nature-based Intervention Condition: Roots and Shoots (Experimental): The intervention condition, Roots and Shoots, consists of a printed, self-help guidebook that incorporates weekly, evidence-based activities with the aim to improve mental wellbeing. The intervention is a short, four week course for improving low wellbeing and is informed by psychological theory, clinical psychology therapeutic principles and environmental psychology.
  Interventions: Behavioral: Roots and Shoots
- Waiting list Control Condition (Active Comparator): Participants in the waiting list control group will complete the assessments at the three time points: baseline (T0), at a 2-weeks (T1) and post-intervention (T2). At this point control condition participants will be offered the intervention and will receive a copy of the Roots and Shoots guidebook in the post and will be provided with full access to the additional online resources.
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: Roots and Shoots — Four-week intervention involving a self-help guidebook to improve mental wellbeing.
  Arms: The Nature-based Intervention Condition: Roots and Shoots
Behavioral: Waiting list — Four-week waiting list period involving treatment as usual.
  Arms: Waiting list Control Condition

SUMMARY:
The goal of this pilot randomised controlled trial is to test the feasibility of a brief nature-based self-help psychological intervention for low mental wellbeing. The investigators want to learn whether the intervention is likely to help improve mental wellbeing and whether it is acceptable to participants. Participants will be members of the public in the United Kingdom (UK) with low mental wellbeing and the intervention lasts for four weeks.

The main questions it aims to answer are:

Will participants' mental wellbeing improve after the intervention, relative to participants in a waiting list arm.

Will participants find the intervention useful and acceptable to do?

Participants will:

Complete baseline questionnaires on demographic information and on several areas linked to wellbeing.

Complete further questionnaires on wellbeing after 2 weeks and 4 weeks. Complete a questionnaire on their experience of the intervention at 4 weeks. Receive and complete a self-guided booklet and link to a webspace to complete activities that are informed by psychological principles.

Receive the intervention after four weeks if they were allocated to the waiting list arm first.

DETAILED DESCRIPTION:
This study tests a brief nature-based psychological intervention for low mental wellbeing. This is a parallel groups waiting list control pilot randomised controlled trial (RCT). This a United Kingdom (UK) based pilot study and has the primary aim of assessing the acceptability and feasibility of the intervention. The pilot will assess the potential for the intervention to improve mental wellbeing but the efficacy of the intervention will be formally tested in a future powered RCT.

This RCT will compare a novel self-help guidebook called 'Roots and Shoots', which was designed to deliver a nature-based intervention for improving low wellbeing, against a waiting list control arm. Eligible participants will be randomly allocated to trial arm (1:1) using random permuted blocks, using the online randomisation service sealedenvelope.com. This is an automated process that ensures randomisation is not influenced by the researchers and prevents selection bias. At baseline (T0), 2-weeks (T1), and 4-weeks (T2) self-report assessments will be collected remotely using the online survey platform, Qualtrics®. Ethical approval was granted by the University of Exeter Psychology Ethics Committee prior to starting the study (Application ID: 5412277).

Participants will be recruited through opportunity sampling using recruitment methods including social media (e.g. Facebook, X), emails, newsletters and printed posters. Participants will be signposted to a brief screening survey in the first instance to check the eligibility criteria. Eligible participants will be contacted via email by a member of the research team to notify them of their eligibility status and confirm their availability to participate in the study. Following confirmation, participants will then be randomly assigned (1:1) to receive the intervention or be placed on a waiting list. Participants will be informed of this outcome by email. Given the nature of the intervention and study design, blinding of the participants is not possible. Participants will receive and read the participant information sheet (PIS) and provide informed consent before commencing the study. Once informed consent has been obtained, all participants will complete a series of baseline measures (T0) prior to starting the intervention or waiting list period. Following receipt of the guidebook, sent to the participant's postal address, participants assigned to the intervention group will be asked to complete the weekly activities and engage with additional online resources housed on the companion website (rowantree.uk).

All participants will be asked to complete a battery of measures at a 2-week interval (T1) and immediate post-intervention, at week 4 (T2). Participants in both the intervention and waiting list control group will complete the same set of online questionnaires at all three timepoints (T0, T1, T2), with the exception of additional feasibility and acceptability questions included in the final survey (T2) for participants in the intervention arm. All measures will be presented to participants in a fixed order and housed in the online distribution platform Qualtrics®. After completion of final survey (at 4-weeks) all participants will receive debrief information which includes the study aims, researcher contact details and signposting for further support and mental health services.

Trial Arms

The Nature-based Intervention: Roots and Shoots

The intervention, Roots and Shoots, consists of a printed, self-help guidebook that covers six main section and includes weekly, evidence-based activities, as well as additional online components. Designed as a short, four week course for improving low wellbeing, the guidebook incorporates elements of environmental psychology (e.g. forest bathing) with techniques and exercises informed by several psychological therapies and traditions. In the first section participants are provided with a comprehensive introduction to the course including nature and wellbeing psychoeducation. This is consistent with research that has highlighted the benefits of psychoeducation as an effective therapeutic approach for improving low mood in individuals with depression. The following four sections guide participants through a set of weekly activities including a habit tracker, psychological coping tool, nature contact tracker, mood and nature connection monitoring and a reflective writing exercise. The rationale for the weekly exercises was informed by behavioural activation principles, mindfulness, cultivation of habits, self-tracking of mood, nature exposure, compassion focused therapy and acceptance and commitment therapy techniques. Throughout Roots and Shoots participants will be signposted to an online webspace where they had access to additional digital resources including nature videos, meditations and breathing exercises. These activities draw on evidence showing the beneficial effects of virtual nature exposure, guided imagery, brief nature-based meditation and guided breathwork. Participants are also encouraged to reflect on their time spent engaging with nature and the guidebook activities.

Waiting list Control

Participants in the waiting list control arm will complete the assessments at the three time points: baseline (T0), at a 2-weeks (T1) and post-intervention (T2). At this point control arm participants will be offered the intervention and will receive a copy of the Roots and Shoots guidebook in the post and will be provided with full access to the additional online resources.

Analyses

Because this is a pilot RCT and is not designed to test the efficacy of the intervention, the primary focus will be on the feasibility and acceptability of the intervention. To this end the investigators will report on the feasibility of the intervention including recruitment to target, and proportion of participants returning the assessment surveys. The investigators will report the simple descriptive statistics on the feasibility and acceptability questions, as well as for the psychometric measures. In the analysis the investigators will follow the principle of intention to treat (ITT). That is, the investigators will not excluding any participants based on their level of engagement with the intervention. The investigators do not plan to remove outliers from any analysis.

The investigators will report the relative change in mean scores on the primary and secondary outcomes. The investigators will primarily report on mean differences, effect sizes and confidence intervals, not p-values. The investigators therefore will not be applying correction for multiple comparisons. No power calculation is required for this pilot study. The investigators will report means, standard deviations and 95% confidence intervals for the psychometric measures and report Hedge's g for estimates of effect size. To assist in the design of a potential future fully powered RCT, the investigators will carry out supplementary analyses. The investigators will carry out repeated measures analyses on the outcomes using mixed models or a general linear model. The investigators will also calculate Clinically Significant Change (CSC) to help assess the clinical significance of any improvement measured in the outcomes. The investigators will explore any clinical change on outcomes using graphs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must score 22 or less on the SWEMWBS scale-indicating low wellbeing-to facilitate clearer assessment of the intervention's consequence on such a measure.
* Participants must be 18+ to take part in the study,
* Participants must have sufficient understanding of the English language, to be able to fully comprehend the measures and intervention tasks, which at present are limited in translation due to methodological constraints.

Exclusion Criteria:

* Visual or auditory impairments that may impede full engagement with the intervention.
* Receiving formal psychological therapy in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2024-06-02 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Short Warwick Edinburgh Mental Wellbeing Scale (SWEMWBS). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Short Warwick Edinburgh Mental Wellbeing Scale (SWEMWBS) is a 7-item unidimensional self-report measure that captures social, eudaimonic and hedonic dimensions of mental wellbeing. Scores range from 7 to 35 and higher scores indicate higher positive mental wellbeing.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-8). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Patient Health Questionnaire (PHQ-8) is an 8-item diagnostic tool and measure used for assessing the severity of depressive symptoms. Scores range from 0 to 24 and higher scores indicate higher severity of depressive symptoms.
Generalised Anxiety Disorder (GAD-7). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Generalised Anxiety Disorder (GAD-7) is a 7-item measure that assesses anxious symptoms during the past 2 weeks. Scores range from 0 to 27 and higher scores indicate higher severity of anxiety symptoms.
Perceived Stress Scale (PSS4). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Perceived Stress Scale (PSS4) is a four-item scale measuring perceived psychological stress in the last month. Scores range from 0 to 16 and higher scores indicate higher levels of perceived stress.
Ruminative Response Styles (RRS). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Ruminative Response Styles (RRS) aims to measure ruminative tendency in response to low mood. The short version of the RRS is comprised of ten items, with two subscales for brooding and reflection. The investigators use only the Brooding subscale, consisting of five items, in this pilot. Scores range from 5 to 20 and higher scores indicate higher levels of rumination.
Five Factor Mindfulness Questionnaire (FFMQ15). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Five Factor Mindfulness Questionnaire (FFMQ15) is a 15-item measure that assesses five aspects of mindfulness including observing, describing, acting with awareness, non-judging and non-reactivity to inner experience. Scores range from 1 to 75 and higher scores indicate higher levels of mindfulness.
Jenkins Sleep Scale (JSS). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Jenkins Sleep Scale (JSS) measures common sleep disturbances symptoms seen in the general population, it contains four items that assess sleep problems over the past month. Scores range from 0 to 20 and higher scores indicate more sleep problems.
The Nature Relatedness Questionnaire (NR6). | T0 (baseline), T1 (2 weeks) and T2 (4 weeks).
  The Nature Relatedness Scale (NR6) is a six-item scale measuring the individual's sense of connection with the natural environment. Scores range from 6 to 35 and higher scores indicate stronger connectedness to nature.
Acceptability and feasibility questions | T2 (4 weeks).
  Please indicate approximately how many days of the guidebook you completed? The guidebook activities were easy to do. The guidebook was easy to follow. The online activities were easy to do. The online activities were easy to follow. I would like the intervention to be longer than 4 weeks. 4 weeks was about the right length for the intervention. I would like the Intervention to be shorter than 4 weeks. Overall I enjoyed doing the Programme. I would come back and use the guidebook again in the future. The Roots & Shoots Programme was helpful in improving my wellbeing. I would recommend the Roots & Shoots Programme to a friend. The information in the guidebook was helpful. The habit wheel was helpful. The habit and mood tracker was helpful. The expressive writing was helpful. The honeycomb challenge was helpful. The coping tool was helpful. I found the nature videos helpful. I found the meditations helpful. I found the breathing exercises helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Owens, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bratman GN, Anderson CB, Berman MG, Cochran B, de Vries S, Flanders J, Folke C, Frumkin H, Gross JJ, Hartig T, Kahn PH Jr, Kuo M, Lawler JJ, Levin PS, Lindahl T, Meyer-Lindenberg A, Mitchell R, Ouyang Z, Roe J, Scarlett L, Smith JR, van den Bosch M, Wheeler BW, White MP, Zheng H, Daily GC. Nature and mental health: An ecosystem service perspective. Sci Adv. 2019 Jul 24;5(7):eaax0903. doi: 10.1126/sciadv.aax0903. eCollection 2019 Jul. PMID 31355340
- [Background] Fincham GW, Strauss C, Montero-Marin J, Cavanagh K. Effect of breathwork on stress and mental health: A meta-analysis of randomised-controlled trials. Sci Rep. 2023 Jan 9;13(1):432. doi: 10.1038/s41598-022-27247-y. PMID 36624160
- [Background] Owens M, Bunce H. The effect of brief exposure to virtual nature on mental wellbeing in adolescents. Sci Rep. 2023 Oct 18;13(1):17769. doi: 10.1038/s41598-023-44717-z. PMID 37853074
- [Background] Owens M, Bunce HLI. Nature-Based Meditation, Rumination and Mental Wellbeing. Int J Environ Res Public Health. 2022 Jul 26;19(15):9118. doi: 10.3390/ijerph19159118. PMID 35897493
- [Background] Tursi MF, Baes Cv, Camacho FR, Tofoli SM, Juruena MF. Effectiveness of psychoeducation for depression: a systematic review. Aust N Z J Psychiatry. 2013 Nov;47(11):1019-31. doi: 10.1177/0004867413491154. Epub 2013 Jun 5. PMID 23739312
- [Background] Uphoff E, Ekers D, Robertson L, Dawson S, Sanger E, South E, Samaan Z, Richards D, Meader N, Churchill R. Behavioural activation therapy for depression in adults. Cochrane Database Syst Rev. 2020 Jul 6;7(7):CD013305. doi: 10.1002/14651858.CD013305.pub2. PMID 32628293
- [Background] van der Watt ASJ, Odendaal W, Louw K, Seedat S. Distant mood monitoring for depressive and bipolar disorders: a systematic review. BMC Psychiatry. 2020 Jul 22;20(1):383. doi: 10.1186/s12888-020-02782-y. PMID 32698802
- See also: Study group and participant webspace. — http://rowantree.uk